CLINICAL TRIAL: NCT03666468
Title: Gaming for Medical Education Research Program: An Investigator-blinded, Randomised Controlled Trial on Serious Games for Doctors, Nurses and Students.
Brief Title: The Gaming for Medical Education Research (G4MER) Program
Acronym: G4MER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Dr Michael Coffey, Principal Investigator, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HC17160-LNR/17/SCHN/194
Record Dates: First submitted 2018-08-14; First posted 2018-09-11 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Education, Medical

STUDY DESIGN:
Intervention Model Description: 3 groups
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PlayMed (Experimental): PlayMed, a highly immersive role-playing computer game
  - Focus on Paediatric Asthma and Seizure management
  Interventions: Other: PlayMed
- Online Package (OP) (Active Comparator): Online package (OP) of NSW Health Guidelines
  - Focus on Paediatric Asthma and Seizure management
  Interventions: Other: Online Package
- Paper Guidelines (Placebo Comparator): Paper NSW Health Guidelines
  - Focus on Paediatric Asthma and Seizure management
  Interventions: Other: Paper Guidelines

INTERVENTIONS:
Other: PlayMed — A highly immersive role-playing computer game focused on Paediatric Asthma and Seizure management
  Arms: PlayMed
Other: Online Package — Online package (OP) of NSW Health Guidelines focused on Paediatric Asthma and Seizure management
  Arms: Online Package (OP)
Other: Paper Guidelines — Paper NSW Health Guideline focused on Paediatric Asthma and Seizure management
  Arms: Paper Guidelines

SUMMARY:
The "G4MER" Program aims to investigate whether serious games add value to medical education in comparison to an online learning package or clinical practice guidelines. The investigators will perform a series of investigator-blinded randomised control trials on doctors, nurses, and medical students at Sydney Children's Hospital. Participants will be given access to their randomly allocated intervention for 8 weeks or 5 days, and will be assessed using multiple choice questions (MCQ) and two observed structure clinical examination (OSCE) stations. Participant attitudes will also be assessed through a mixed-methods questionnaire.

DETAILED DESCRIPTION:
The "G4MER" Program aims to perform a series of randomised control trials on different groups at Sydney Children's Hospital:

1. Study 1A (Formerly titled "Serious Games in Medical Education - a Randomised Control Trial") is already underway and involves Phase 3 medical students at UNSW having 8 weeks access to the game, an Online Package (OP) or NSW State Guidelines on Asthma and Seizure management. Students are then assessed using multiple choice questions (MCQ) and two observed structure clinical examination (OSCE) stations (detailed below).
2. Study 1B is also a randomised control trial similar in design to Study 1A, however it will involve doctors and nurses employed at Sydney Children's Hospital. PlayMed will be compared against the HETI Learning Path Paediatric Clinical Practice Guidelines (Online Package for staff).
3. Studies 2A and 2B are identical to Studies 1A and 1B respectively except participants will have 2 hours access to their educational tool. Participants will then immediately undergo the same assessment using multiple choice questions (MCQ) and two observed structure clinical examination (OSCE) stations The proposed study designs are all blinded randomised control trials. Participants may only be involved in Study 1 or Study 2, not both.

Administration

Studies 1A and 1B Participants allocated to the game and to the OP will be given the appropriate access for 8 weeks (instructions provided in the study envelope). Participants allocated to the guidelines will receive a print-out of the guidelines. Participants will be encouraged to engage with their additional educational tool as often as they wish during their eight weeks. In the 8th last week participants will have their knowledge and clinical performance assessed as outlined below.

Studies 2A and 2B Participants allocated to the game, OP and guidelines will be given 2 hours to utilise their assigned teaching tool. Two hours was selected as an appropriate time-frame in which participants would be able complete all cases of the game or online package, or read through the guidelines. Furthermore, it was chosen as it is more pragmatic and better at assessing short-term retention. Computers will be provided for participants to access the game and OP. The guidelines will be printed for participants to read. Participants will then immediately have their knowledge and clinical performance assess as outlined below.

Assessment

Studies 1A, 1B, 2A and 2B Participants will be assessed for knowledge acquisition and clinical performance. Participant knowledge will be assessed using 10 multiple choice questions (MCQ). Participant clinical skills will be assessed via an observed structured clinical examination (OSCE) administered in the simulation laboratory (immediately after the knowledge test); participants will be tested across two clinical scenarios. Strict marking criteria will be used to ensure standardisation.

ELIGIBILITY:
Inclusion Criteria:

* Studies 1A and 2A Phase 2 or 3 medical students at UNSW who are enrolled in the Children's Health Course will be eligible
* Studies 1B and 2B Doctors and nurses employed at Sydney Children's Hospital.

Exclusion Criteria:

* Studies 1A and 2A Medical students not actively enrolled at UNSW
* Studies 1B and 2B Doctors and nurses not actively employed at Sydney Children's Hospital.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2017-07-03 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Multiple choice quiz score | Post-intervention assessment; 8 weeks (Study 1A and 1B) or 2 hours (Study 2A and 2B).
  A paper-based assessment using multiple choice questions designed to test knowledge acquisition for asthma and seizure management. For Studies 1A and 1B, scale 0 to 10, higher is better performance. Studies 2A and 2B, scale from 0 to 15, higher is better.
Asthma observed structured clinical examination (OSCE) score | Post-intervention assessment; 8 weeks (Study 1A and 1B) or 2 hours (Study 2A and 2B).
  An OSCE administered in a high-fidelity simulation lab. A child with an exacerbation of asthma will be presented and the management required will need to be implemented by the participant. For Studies 1A and 1B, subscale from 0 to 15, higher is better, with scores summed with Outcome 3. Studies 2A and 2B, subscale from 0 to 25, higher is better, with scores summed with Outcome 3.
Seizure observed structured clinical examination (OSCE) scoresimulation lab) | Post-intervention assessment; 8 weeks (Study 1A and 1B) or 2 hours (Study 2A and 2B).
  An OSCE administered in a high-fidelity simulation lab. A child with a seizure will be presented and the management required will need to be implemented by the participant. For Studies 1A and 1B, subscale from 0 to 15, higher is better, with scores summed with Outcome 3. Studies 2A and 2B, subscale from 0 to 25, higher is better, with scores summed with Outcome 2.

SECONDARY OUTCOMES:
Participant attitudes towards educational intervention | Post-intervention assessment; 8 weeks (Study 1A and 1B) or 2 hours (Study 2A and 2B).
  Mixed-methods analysis survey. 5-point Likert scale from "Strongly Agree" to "Strongly Disagree".
Time to specific actions in OSCE scenarios | Post-intervention assessment; 8 weeks (Study 1A and 1B) or 2 hours (Study 2A and 2B).
  E.g. calling for help, oxygen supplementation, salbutamol, anti-epileptic drug
Anti-epileptic medication(s) administered at correct time during OSCE scenario | Post-intervention assessment; 8 weeks (Study 1A and 1B) or 2 hours (Study 2A and 2B).
  E.g. Midazolam or diazepam correctly administered at 5 minutes of seizure activity (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Coffey, BMed MD, Principal Investigator — The University of New South Wales
Locations (1):
- Sydney Children's Hospital, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT03666468/Prot_SAP_000.pdf